CLINICAL TRIAL: NCT03379129
Title: Validation of Family-Administered Delirium Detection Tools for the Identification of Delirium in Critically Ill Patients
Brief Title: Family ICU Delirium Detection Study
Acronym: FIDDS
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Other Study IDs: REB-16-2060
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2017-11

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the validity, reliability, and acceptability of employing family-administered delirium detection tools in the critically ill. The ultimate goal of this project is to improve the care of critically ill patients by creating valid, earlier, and patient and family-centered prevention, recognition, and management of delirium.

DETAILED DESCRIPTION:
Delirium is a major problem in critically ill patients, affecting almost half of this population. Delirium is associated with substantial persistent impaired cognition and psychiatric comorbidity, attributable mortality, and increased healthcare costs. Family members of critically ill patients are also at risk for developing adverse consequences including anxiety and depression. One strategy that may help both patients and families is to engage family members in the detection of delirium. The Facilitated Sensemaking model (of family member/patient engagement in critical care) is the theoretical framework underpinning the proposed work. Facilitated Sensemaking engages families by providing opportunities to participate in communication, decision-making, and bedside care, with the understanding that a sense of purpose derived from active participation in care can serve as a protective mechanism to reduce stress-related complications among families of critically ill patients, known as Post-Intensive Care Syndrome-Family. Family delirium detection may result in earlier and more accurate recognition of delirium and meaningful family involvement, and therein the potential for better patient and family outcomes. Family-administered tools to measure delirium exist, but they have not been explored in the intensive care unit (ICU) context; the ICU is unique in terms of the patient population served and the invasiveness of therapies employed. We propose to evaluate the validity and reliability of using family-administered tools to detect delirium in critically ill patients and to explore perceptions and experiences of family members' participation in the detection of delirium.

Aim 1: To assess the validity and reliability of the Family Confusion Assessment Method (FAM-CAM) and Sour Seven to detect delirium in critically ill patients (Phase 1).

Aim 2: To explore stakeholder (former ICU patients and family members, nurse, physician) perceptions and experiences of family-administered delirium detection in critically ill patients (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Richmond Agitation Sedation Scale (RASS) ≥-3
* able to communicate with study team (understand English, no significant hearing impairment)
* located in ICU

Exclusion Criteria:

* Significant primary direct brain injury with a Glasgow Coma Score (GCS) of <9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and family members in the largest adult ICU in Calgary, Alberta (Foothills Medical Centre, FMC) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Eleven item Family Confusion Assessment Method (FAM-CAM) family caregiver administered delirium detection tool | up to 5 days
  To be completed by a family caregiver once per day. The FAM-CAM is considered positive if acute onset (Question 1,10) or fluctuating course (question 9) AND inattention (question 2) AND either disorganized thinking (question 3,5,6) or altered consciousness (question 4) are present. This tool will be validated against intensive care unit (ICU) registered nurse (RN) reference standard ratings for delirium.
Seven item Sour Seven family caregiver administered delirium detection tool | up to 5 days
  To be completed by a family caregiver once per day. Possible delirium is indicated by a score of 4 and higher. Any score of 9 or higher indicates delirium is present. This tool will be validated against ICU RN reference standard ratings for delirium.

SECONDARY OUTCOMES:
Seven item General Anxiety Disorder (GAD-7) questionnaire to detect signs of anxiety in the family caregivers at the bedside | up to 5 days
  Scores of 5, 10 and 15 indicate signs of mild, moderate and sever anxiety, respectively
Nine item Patient Health Questionnaire (PHQ-9) questionnaire to detect signs of depression in the family caregiver at the bedside | up to 5 days
  Depression severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten M Fiest, PhD, Principal Investigator — University of Calgary; Henry T Stelfox, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital ICU, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Poulin TG, Krewulak KD, Rosgen BK, Stelfox HT, Fiest KM, Moss SJ. The impact of patient delirium in the intensive care unit: patterns of anxiety symptoms in family caregivers. BMC Health Serv Res. 2021 Nov 5;21(1):1202. doi: 10.1186/s12913-021-07218-1. PMID 34740349
- [Derived] Parsons Leigh J, Krewulak KD, Zepeda N, Farrier CE, Spence KL, Davidson JE, Stelfox HT, Fiest KM. Patients, family members and providers perceive family-administered delirium detection tools in the adult ICU as feasible and of value to patient care and family member coping: a qualitative focus group study. Can J Anaesth. 2021 Mar;68(3):358-366. doi: 10.1007/s12630-020-01866-3. Epub 2020 Nov 18. PMID 33210217
- [Derived] Krewulak KD, Sept BG, Stelfox HT, Ely EW, Davidson JE, Ismail Z, Fiest KM. Feasibility and acceptability of family administration of delirium detection tools in the intensive care unit: a patient-oriented pilot study. CMAJ Open. 2019 Apr 26;7(2):E294-E299. doi: 10.9778/cmajo.20180123. Print 2019 Apr-Jun. PMID 31028053